CLINICAL TRIAL: NCT07217951
Title: Assessing the Feasibility of Multi-modal Biosensing for Monitoring Mobility and Cognition in Older Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01AG091766 (NIH); R01AG091766 (NIH)
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Chronic Stress; Systemic Inflammation; Mobility and Independence
Keywords: wearable sensors; older adults; aging; mobility; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults: Adults aged 65 or older
  Interventions: Device: Eutectogel Sensors and Microneedle Patches

INTERVENTIONS:
Device: Eutectogel Sensors and Microneedle Patches — Eutectogel Sensors:
  While the exact eutectogel formulation in this study has not been previously tested in humans, similar eutectogel-based materials have been employed in wearable biosensing devices with human participants. These systems are typically composed of biocompatible matrices such as gelatin or polyacrylamide combined with deep eutectic solvents (DES) to improve ionic conductivity and flexibility.
  Microneedle Patches:
  The microneedle patch in this study is composed of poly(acrylic acid)/gelatin methacryloyl (PAA/GelMA), gelatin/oxidized pectin (Gelatin/OxP), and methacrylated hyaluronic acid/maleic anhydride (MeHA/MA). Although the integrated use of these specific compositions has not yet been evaluated in humans, the materials themselves, as well as similar microneedle architectures, have been thoroughly investigated in vivo and even in clinical trials.

SUMMARY:
Current health devices often overlook older users, who may face both health challenges and technology barriers. We are investigating the feasibility of wearable sensors to track posture, heart rate, and breathing, alongside a microneedle patch that collect body fluids to measure stress and inflammation markers. By combining this data, we aim to create an easy to use system that supports personalized, at home health monitoring for older adults.

DETAILED DESCRIPTION:
Devices capable of measuring, interpreting, and providing guidance based on a range of biosignals have significantly broadened the access to health information. Nevertheless, the majority of these platforms are designed for a demographic already proficient in technology, thereby excluding older adults, a group facing unique health challenges and often experiencing technological apprehension. To address this disparity, this study aims to demonstrate the feasibility of employing a wearable eutectogel-sensor patch system to monitor and analyze posture, movement, heart rate, and respiration of older adults within their natural living environments. Furthermore, investigators seek to develop algorithms that correlate these real-time data streams with physical and cognitive performance outcomes. Concurrently, they will investigate the feasibility of employing hydrogel microneedle patches for the passive collection of interstitial fluid (ISF) to measure key biomarkers associated with stress and inflammation, specifically cortisol, dopamine, and C-reactive protein (CRP). These biomarkers serve as critical indicators of physiological stress, mood regulation, and systemic inflammation, which are closely associated with cognitive decline, frailty, and diminished quality of life in the aging population. Eutectogel sensor patches are flexible, breathable, inconspicuous, and designed for long-term wear. They can be positioned strategically to provide direct, continuous, real-time monitoring of posture, motion, heart rate, and respiration. We now propose to determine the feasibility of using a eutectogel sensor patch system to continuously collect posture, motion, heart rate, and respiration data in free-living older adults. Investigators will secondly assess the feasibility of measuring dopamine, cortisol, and CRP from ISF collected with a microneedle patch and correlate them with the same analytes measured in saliva. These analytes were selected due to their relevance in detecting chronic stress and systemic inflammation-conditions that are highly prevalent and often underdiagnosed in the aging population. The research objectives are significant because they aim to bridge the technological and demographic gap through a combined sensing system that enables seamless and meaningful health monitoring in real-world settings.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 or older
2. Expressed willingness to participate.
3. Able to give written informed consent
4. Able to operate a smartphone and complete surveys

Exclusion Criteria:

1. Reliance on assistive walking devices
2. Inability to operate a smartphone
3. Unable to complete surveys
4. Unable to give written informed consent
5. Younger than 65 years old
6. Known skin allergies to kinesiology tape (KT tape)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults aged 65 and older.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Subtle biomechanical signals and interstitial fluid with key biomarkers. | From enrollment to end of study period at 8 days.
  We propose the use of eutectogel-based strain sensors as a soft, conformable platform for capturing subtle biomechanical signals, including posture shifts, respiratory motion, and joint movements. These gels offer unique advantages in comfort and stretchability that make them ideal for long-term use by older adults. Complementing this, we integrate hydrogel-based microneedle patches for the continuous and minimally invasive collection of interstitial fluid to measure key biomarkers: cortisol and dopamine (using the PAA/GelMA microneedle-dPAD system) and C-reactive protein (via the Gelatin/OxP microneedle µPAD platform). These biomarkers are critically relevant to monitoring stress, inflammation, and mental health-all major contributors to declining independence in aging populations. By applying machine learning methods to passively interpret this multimodal dataset, our approach addresses the unmet need for integrated, unobtrusive health monitoring systems tailored to the aging popula

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Sonkusale, PhD, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Dongiovanni P, Meroni M, Casati S, Goldoni R, Thomaz DV, Kehr NS, Galimberti D, Del Fabbro M, Tartaglia GM. Salivary biomarkers: novel noninvasive tools to diagnose chronic inflammation. Int J Oral Sci. 2023 Jun 29;15(1):27. doi: 10.1038/s41368-023-00231-6. PMID 37386003
- [Background] Wu Z, Qiao Z, Chen S, et al. Interstitial fluid-based wearable biosensors for minimally invasive healthcare and biomedical applications. Communications Materials. 2024;5(1):33. 10.1038/s43246-024-00468-6,
- [Background] Cheng KC, Aeron S, Hughes MC, Miller EL. Nonparametric and Regularized Dynamical Wasserstein Barycenters for Sequential Observations. IEEE Transactions on Signal Processing. 2022;71:3164-3178.
- [Background] Cheng K, Aeron S, Hughes MC, Miller EL. Dynamical Wasserstein barycenters for time-series modeling. Advances in Neural Information Processing Systems. 2021;34:27991-28003
- [Background] Zhang H, Miller EL, Abriola LM. Manifold regression for subsurface contaminant characterization based on sparse concentration data. Paper presented at: 2014 IEEE Geoscience and Remote Sensing Symposium; 13-18 July 2014, 2014.
- [Background] Bhattarai KR, Kim HR, Chae HJ. Compliance with Saliva Collection Protocol in Healthy Volunteers: Strategies for Managing Risk and Errors. Int J Med Sci. 2018 May 22;15(8):823-831. doi: 10.7150/ijms.25146. eCollection 2018. PMID 30008593
- [Background] Gupta S, Nayak MT, Sunitha JD, Dawar G, Sinha N, Rallan NS. Correlation of salivary glucose level with blood glucose level in diabetes mellitus. J Oral Maxillofac Pathol. 2017 Sep-Dec;21(3):334-339. doi: 10.4103/jomfp.JOMFP_222_15. PMID 29391704
- [Background] Iijima H, Shimoura K, Eguchi R, Aoyama T, Takahashi M. Concurrent validity and measurement error of stair climb test in people with pre-radiographic to mild knee osteoarthritis. Gait Posture. 2019 Feb;68:335-339. doi: 10.1016/j.gaitpost.2018.12.014. Epub 2018 Dec 10. PMID 30576977
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Gelatin Food additive and GRAS regulations. U.S. Food and Drug Administration; 2025.
- [Background] 184.1724 Sodium Alginate. Code of Federal Regulations Title 21.
- [Background] CELLULOSE, MICROCRYSTALLINE. U.S. Food and Drug Administration; 2025
- [Background] Master H, Coleman G, Dobson F, Bennell K, Hinman RS, Jakiela JT, White DK. A Narrative Review on Measurement Properties of Fixed-distance Walk Tests Up to 40 Meters for Adults With Knee Osteoarthritis. J Rheumatol. 2021 May;48(5):638-647. doi: 10.3899/jrheum.200771. Epub 2020 Oct 15. PMID 33060316
- [Background] 182.1320 Glycerin. Code of Federal Regulations Title 21, Environmental Protection Agency; 2025
- [Background] Zhang J, Li H, Albakr L, Zhang Y, Lu A, Chen W, Shao T, Zhu L, Yuan H, Yang G, Wheate NJ, Kang L, Wu C. Microneedle-enabled therapeutics delivery and biosensing in clinical trials. J Control Release. 2023 Aug;360:687-704. doi: 10.1016/j.jconrel.2023.07.023. Epub 2023 Jul 19. PMID 37442203
- [Background] Zhu J, Zhou X, Kim HJ, et al. Gelatin Methacryloyl Microneedle Patches for Minimally Invasive Extraction of Skin Interstitial Fluid. Small. 2020;16(16):e1905910. PMC7182487. 9. Chang H, Zheng M, Yu X, et al. A Swellable Microneedle Patch to Rapidly Extract Skin Interstitial Fluid for Timely Metabolic Analysis. Adv Mater. 2017;29(37). 10.1002/adma.201702243
- [Background] Long W, George Joy J, Lee SJ, Kim JC. Collagen- and Hyaluronic Acid-Based Microneedles With Thiolated Pectin for Redox-Responsive Drug Delivery. J Biomed Mater Res A. 2025 Apr;113(4):e37903. doi: 10.1002/jbm.a.37903. PMID 40156176
- [Background] Shu Y, Qi Y, Zou Y, Huang Y, Chen J, Li J, Chen L, Zhu X. A gelatin microneedles featuring antibacterial and reactive oxygen species scavenging properties for treating Vibrio vulnificus-infected wounds. Int J Biol Macromol. 2025 May;309(Pt 1):142640. doi: 10.1016/j.ijbiomac.2025.142640. Epub 2025 Mar 28. PMID 40158599
- [Background] Liu D, Wang S, Wang H, Zhang Z, Wang H. A flexible, stretchable and wearable strain sensor based on physical eutectogels for deep learning-assisted motion identification. J Mater Chem B. 2024 Jun 27;12(25):6102-6116. doi: 10.1039/d4tb00809j. PMID 38836422
- [Background] Lu Q, Li H, Tan Z. Zwitterionic Eutectogel-Based Wearable Strain Sensor with Superior Stretchability, Self-Healing, Self-Adhesion, and Wide Temperature Tolerance. ACS Appl Mater Interfaces. 2023 Jul 19;15(28):34055-34063. doi: 10.1021/acsami.3c05848. Epub 2023 Jul 6. PMID 37410953
- [Background] Wang Y, Zhou W, Shen C, Jiang G, Yang C. Flexible and printable integrated biosensors for monitoring sweat and skin condition. Anal Biochem. 2023 Jan 15;661:114985. doi: 10.1016/j.ab.2022.114985. Epub 2022 Nov 19. PMID 36414087
- [Background] Qin H, Owyeung RE, Sonkusale SR, Panzer MJ. Highly stretchable and nonvolatile gelatin-supported deep eutectic solvent gel electrolyte-based ionic skins for strain and pressure sensing. Journal of Materials Chemistry C. 2019;7(3):601-608. 10.1039/C8TC05918G
- [Background] Wei Z, Jia L, Yu J, Xu H, Guo X, Xiang T, Zhou S. Environmentally tolerant multifunctional eutectogel for highly sensitive wearable sensors. Mater Horiz. 2025 Apr 14;12(8):2604-2618. doi: 10.1039/d4mh01665c. PMID 39806946